CLINICAL TRIAL: NCT00259129
Title: Effect of BAY 43-9006 (Sorafenib) on Cardiovascular Safety Parameters in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 100561
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 400 mg twice a day (bid) (2 x 200 mg tablets)

SUMMARY:
This is an open-label, non-randomized Phase I study of sorafenib 400 mg bid (2 x 200 mg tablets) in cancer patients. The primary objective of the study is to evaluate the effect of sorafenib on cardiovascular safety parameters. The secondary objectives are to evaluate the safety, pharmacokinetics, and anti-tumor activity of sorafenib in cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory solid cancer for which curative or palliative measures have failed or patients for whom standard treatment is considered ineffective or intolerable
* Histological or cytological documentation of cancer is required
* Patients with at least one evaluable lesion. Lesions must be evaluated by Computed Tomography (CT) scan or Magnetic Resonance Imaging (MRI)
* Life expectancy of at least 12 weeks
* Left ventricular ejection fraction (LVEF) >=45 % as assessed at the Baseline Multiple Gated Acquisition (MUGA) scan
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to dosing:

  * Hemoglobin > 9.0 g/dL
  * Absolute neutrophil count (ANC) > 1,500/mm3
  * Platelet count >=100,000/dL
  * Total bilirubin <=1.5 times the upper limit of normal
  * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) <=2.5 x upper limit of normal, except if there is metastatic disease to the liver, in which case <=5 x upper limit of normal is acceptable
  * Prothrombin Time-International Normalized Ratio/Partial Thromboplastin Time (PT-INR/PTT) < 1.5 x upper limit of normal. Patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists. For patients on anticoagulation therapy, at least weekly evaluations will be performed until International Normalized Ratio (INR) is stable as defined by the local standard of care
* Serum creatinine <=1.5 x upper limit of normal

Exclusion Criteria:

* Colorectal cancer whether refractory or not
* Supine systolic blood pressure greater than 170 mmHg or diastolic blood pressure greater than 100 mmHg (mean of duplicate readings) at Screening with or without antihypertensives
* Symptomatic metastatic brain or meningeal tumors
* Pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-08; Primary Completion 2007-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Effect of sorafenib on cardiovascular safety parameters | up to 2 months

SECONDARY OUTCOMES:
Pharmacokinetics | after 16 months
Anti-tumor activity | after 10 months
Adverse Event Collection | after 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Boston, Massachusetts
  - San Antonio, Texas

REFERENCES:
- [Result] Tolcher AW, Appleman LJ, Shapiro GI, Mita AC, Cihon F, Mazzu A, Sundaresan PR. A phase I open-label study evaluating the cardiovascular safety of sorafenib in patients with advanced cancer. Cancer Chemother Pharmacol. 2011 Apr;67(4):751-64. doi: 10.1007/s00280-010-1372-3. Epub 2010 Jun 3. PMID 20521052